CLINICAL TRIAL: NCT00002913
Title: PHASE I STUDY OF PACLITAXEL COMBINED WITH TOPOTECAN AND CISPLATIN AND G-CSF IN PATIENTS WITH NEWLY DIAGNOSED ADVANCED OVARIAN EPITHELIAL MALIGNANCIES
Brief Title: Paclitaxel, Cisplatin, and Topotecan With or Without Filgrastim in Treating Patients With Newly Diagnosed Stage III or Stage IV Epithelial Ovarian Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02251; GOG-9602; U10CA027469 (NIH); CDR0000065286 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Brenner Tumor; Ovarian Clear Cell Cystadenocarcinoma; Ovarian Endometrioid Adenocarcinoma; Ovarian Mixed Epithelial Carcinoma; Ovarian Mucinous Cystadenocarcinoma; Ovarian Serous Cystadenocarcinoma; Ovarian Undifferentiated Adenocarcinoma; Stage III Ovarian Epithelial Cancer; Stage IV Ovarian Epithelial Cancer
MeSH Terms: conditions — Brenner Tumor; Carcinoma, Ovarian Epithelial | interventions — Paclitaxel; Taxes; Cisplatin; Topotecan; trioctyl phosphine oxide; Filgrastim; Granulocyte Colony-Stimulating Factor

ARMS (1):
- Treatment (paclitaxel, cisplatin, topotecan hydrochloride) (Experimental): Patients receive paclitaxel IV over 3 hours and cisplatin IV on day 1, followed by topotecan IV over 30 minutes on days 1-3. Patients receive filgrastim (G-CSF) subcutaneously beginning on day 4 and continuing until blood counts recover. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Cohorts of 4-6 patients receive escalating doses of topotecan until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose limiting toxicities.
  Interventions: Drug: paclitaxel; Drug: cisplatin; Drug: topotecan hydrochloride; Biological: filgrastim

INTERVENTIONS:
Drug: paclitaxel — Given IV
  Other Names: Anzatax; Asotax; TAX; Taxol
Drug: cisplatin — Given IV
  Other Names: CACP; CDDP; CPDD; DDP
Drug: topotecan hydrochloride — Given IV
  Other Names: hycamptamine; Hycamtin; SKF S-104864-A; TOPO
Biological: filgrastim — Given SC
  Other Names: G-CSF; Neupogen

SUMMARY:
Phase I trial to study the effectiveness of paclitaxel, cisplatin, and topotecan with or without filgrastim in treating patients who have newly diagnosed stage III or stage IV epithelial ovarian cancer. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Colony-stimulating factors such as filgrastim may increase the number of immune cells found in bone marrow or peripheral blood and may help a person's immune system recover from the side effects of chemotherapy

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated doses of paclitaxel, cisplatin, and topotecan administered together with or without filgrastim (G-CSF) in patients with newly diagnosed advanced ovarian cancer.

II. Describe and quantitate the clinical toxic effects of combination chemotherapy with paclitaxel, cisplatin, and topotecan with or without G-CSF.

III. Assess preliminary evidence of antitumor activity of this combination chemotherapy in these patients.

OUTLINE: This is a dose escalation study of topotecan.

Patients receive paclitaxel IV over 3 hours and cisplatin IV on day 1, followed by topotecan IV over 30 minutes on days 1-3. Patients receive filgrastim (G-CSF) subcutaneously beginning on day 4 and continuing until blood counts recover. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 4-6 patients receive escalating doses of topotecan until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose limiting toxicities.

Patients are followed as clinically indicated.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed epithelial ovarian carcinoma

  * No borderline ovarian carcinoma
  * Stage III/IV disease that has been suboptimally or optimally debulked
* The following histologies are eligible:

  * Adenocarcinoma (unspecified)
  * Mucinous cystadenocarcinoma
  * Clear cell adenocarcinoma
  * Serous cystadenocarcinoma
  * Endometrioid adenocarcinoma
  * Transitional cell carcinoma
  * Malignant Brenner's tumor
  * Undifferentiated carcinoma
  * Mixed epithelial carcinoma
  * Extraovarian papillary serous cystadenocarcinoma
* Measurable or evaluable disease
* Performance status - GOG 0-1
* Enabling completion of at least 2 courses of therapy
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin no greater than 1.5 mg/dL
* Creatinine clearance at least 60 mL/min
* No myocardial infarction within 6 months
* No congestive heart failure
* No unstable or uncontrolled angina
* No history of cardiac arrhythmia requiring anti-arrhythmia medication
* No uncontrolled hypertension
* No hypersensitivity to E. coli-derived drug preparation
* No active infection
* No sensory neuropathy
* No other malignancies within the past 5 years except nonmelanomatous skin cancer
* No prior chemotherapy
* No prior radiotherapy
* Recovered from any recent surgery

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 1996-12; Primary Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Maximally tolerated doses (MTDs) of the combination of paclitaxel, Topotecan, and cisplatin administered without and with G-CSF based on dose-limiting toxicities (DLT) graded according to GOG Common Toxicity Criteria | 3 weeks

SECONDARY OUTCOMES:
Overall survival | Up to 10 years
Progression-free survival | Up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Armstrong, Principal Investigator — Gynecologic Oncology Group
Locations (1):
- Gynecologic Oncology Group of Arizona, Phoenix, Arizona, United States